CLINICAL TRIAL: NCT02005211
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Effect on Biomarkers of AZD3293 in Healthy Japanese Male and Non-Fertile Female Volunteers Including Elderly
Brief Title: A Two-part Single and Multiple Dose Study to Assess the Safety , Pharmacokinetics and Effects of AZD3293 in Healthy Japanese Young and Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D5010C00003
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Japanese Young and Elderly Male and Non-fertile Female Volunteers
Keywords: AZD3293; Healthy volunteers; Young volunteers; Elderly volunteers; Japanese volunteers; Phase 1; Single and multiple ascending dose study
MeSH Terms: interventions — lanabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD3293 (Experimental): AZD3293 will be administered as single dose of an oral solution in Part 1 and single and multiple doses of an oral solution in Part 2. The ascending doses are planned to be 15, 50 and 150 mg for young subjects in Part 1 and 15 and 50 mg for elderly subjects in Part 2. Before proceeding to next dose level, safety, tolerability and pharmacokinetic data from the previous cohort(s) will be evaluated by a Safety Review Committee. Part 2 will start after confirming safety and tolerability in Part 1.
  Interventions: Drug: AZD3293
- Placebo (Placebo Comparator): Placebo given (2 subjects in each cohort)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3293 — Oral solution
  Arms: AZD3293
Drug: Placebo — Oral solution
  Arms: Placebo

SUMMARY:
This study consists of two parts, ie, single dose part with young healthy subjects (Part 1) and single and multiple dose part with elderly healthy subjects (Part 2), to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD3293 following single and multiple ascending dose administration to healthy subjects.

DETAILED DESCRIPTION:
This is a Phase I, randomised, double-blind, placebo-controlled, single centre study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD3293 following single and multiple ascending dose administration to healthy subjects. This study consists of two parts, ie, single dose part with young healthy subjects (Part 1) and single and multiple dose part with elderly healthy subjects (Part 2). The study design allows a gradual escalation of dosage levels between sequential cohorts with safety monitoring to ensure the safety of the healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese elderly and young males and females (of non-childbearing potential)
* Body mass index (BMI) between 17 and 27 kg/m2 and weigh at least 40 kg and no more than 100 kg

Exclusion Criteria:

* Psychiatric disease/condition, GI, renal, hepatic, cardiovascular, psychiatric, or retinal diseases or disorders
* Use of antipsychotic drugs , or chronic use of antidepressant or anxiolytic drugs.
* Frequent use (more than 2 days per week during the last 12 weeks) of tobacco or other nicotine products.
* Neurological disease, including seizures, recent memory impairment, or clinically significant head injury.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Alexander, MD, Study Director — AstraZeneca; Kei Sakamoto, MD, PhD, Principal Investigator — Sugioka Memorial Hospital, Medical Co. LTA
Locations (1):
- Research Site, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects, adult and elderly Japanese vlounteers, male and female (non-fertile); First patient enrolled 24 Dec 2013, last patient completed 29 Jul 2014
Pre-assignment Details: Single Japanese Centre: SAD Part 1: 24 young adult subjects in 3 cohorts of 8, 2 placebo and 6 active AZD3293 dose (15 mg, 50 mg, 150 mg); MAD Part 2:16 elderly subjects in 2 Cohorts of 8, randomized 2 placebo and 6 active dose AZD3293 (15 mg, 50 mg) - Only data on subjests enrolled into cohorts was included in the data base for reporting
Groups:
- Placebo Part 1: Placebo Part 1 - SAD
- AZD3293 15 mg Part 1: AZD3293 15 mg Part 1 - SAD
- AZD3293 50 mg Part 1: AZD3293 50 mg Part 1 - SAD
- AZD3293 150 mg Part 1: AZD3293 150 mg Part 1 - SAD
- AZD3293 15 mg Part 2: AZD3293 15 mg Part 2 -MAD
- AZD3293 50 mg Part 2: AZD3293 50 mg Part 2 - MAD
- Placebo Part 2: Placebo Part 2 - MAD
Period: Part 1 - Cohorts 1-3 Adult Subjects
Arm/Group | Placebo Part 1 | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2 | Placebo Part 2
Started | 6 | 6 | 6 | 6 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 - Elderly Subjects Cohorts 4 & 5
Arm/Group | Placebo Part 1 | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2 | Placebo Part 2
Started | 0 | 0 | 0 | 0 | 6 | 6 | 4
Completed | 0 | 0 | 0 | 0 | 5 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1 - Single Ascending Dose - healthy adults, Part 2 - Multiple Ascending Doses - healthy elderly
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Part 1 | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2 | Placebo Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at study enrollment
  Years
    Young adult | 28.8 (9.1) [20 to 42] | 32.2 (9.7) [22 to 46] | 23.8 (5.0) [21 to 34] | 22.7 (3.3) [20 to 29] | NA (NA) — Elderly | NA (NA) [59 to 70] — Elderly | NA (NA) [56 to 68] — Elderly | 26.9 (7.8) [56 to 71]
    Elderly Adults | NA (NA) — Young | NA (NA) — Young | NA (NA) — Young | NA (NA) — Young | 65.5 (3.8) [59 to 71] | 64.2 (5.0) | 60.5 (5.4) | 63.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 4 | 5 | 3 | 12
  Male | 6 | 6 | 6 | 6 | 2 | 1 | 1 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 40

OUTCOME MEASURES:

1. Secondary Outcome: PK Cmax - Overall Study
Description: Pharmacokinetic maximum concentration
Time Frame: 0, 0.5,1,2,3,4,8,12,24,48 hr single dose, multiple dose does not include 48 hr
Population: Pharmacokinetic
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
ng/mL
  Single dose | 82.5 (20.9) | 395 (24.9) | 1480 (14.4) | 86.6 (31.7) | 395 (38.5)
  MAD -Day 10 steady state | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | 115 (29.7) | 465 (42.2)
  MAD - Day 14 steady state | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | 119 (23.3) | 502 (30.6)

2. Secondary Outcome: PK AUC - Overall Study (SAD & MAD Parts)
Description: Pharmacokintic Area Under the Curve (0 to t)
Time Frame: 0,0.5,1,2,3,4,8,12,24,48 hr single dose, multiple dose does not include 48 hr
Population: healthy Japanese participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.ng/mL
Arm/Group | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
hr.ng/mL
  Single dose | 839 (28.1) | 2810 (17.6) | 10700 (10.1) | 877 (12.5) | 3070 (27.7)
  MAD -Day 10 Steady state | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | 1060 (18.3) | 3540 (37.3)
  MAD -Day 14 Steady state | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | 1030 (12.8) | 3280 (30.4)

3. Secondary Outcome: Biomarker
Description: Biomarker (Abeta 1-40; A beta 1-42) % change from baseline
Time Frame: Pre dose vs Day 14
Population: Pharmacodynamic
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Placebo Part 1 | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2 | Placebo Part 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 4
% change from baseline
  Plasma Abeta(1-40), Day 1 | -9.03 (14.3) | -69.6 (8.36) | -75.8 (6.34) | -62.7 (37.6) | -65.9 (4.54) | -70.2 (3.76) | -7.4 (3.89)
  Plasma Abeta (1-42) Day 1 | 4.80 (9.78) | -58.3 (22.3) | -71.9 (9.74) | -79.4 (4.84) | -73.7 (4.03) | -77.1 (5.31) | 12.4 (16.9)
  Plasma Abeta(1-40) Day 14 | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | -74.7 (5.28) | -77.0 (3.36) | -5.1 (8.56)
  CSF Abeta(1-40) Day 14 | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | -50.4 (7.49) | -76.6 (3.96) | -8.0 (22.7)
  CSF Abeta(1-42) Day 14 | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | -63.2 (9.12) | -79.3 (4.69) | 1.75 (21.9)
  Plasma Abeta(1-42) Day 14 | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | NA (NA) — PART 1 - Single dose | -77.6 (4.73) | -78.6 (4.27) | 15.9 (19.9)

4. Primary Outcome: Safety - Adverse Events
Description: Safety - Number of subjects reporting any adverse events during the study
Time Frame: Day of first dose to follow up
Population: Safety
Measure: Number; unit: Participants
Groups:
- Placebo Part2: Placebo Part 2 - MAD
Arm/Group | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2 | Placebo Part 1 | Placebo Part2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Participants | 1 | 1 | 0 | 2 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 10 days after last dose, for Part 1: 7 to 10 days; for Part 2: 21 to 24 days
Description: Treatment emergent AEs were recorded from day of 1st dose
Arm/Group | Placebo Part 1 | AZD3293 15 mg Part 1 | AZD3293 50 mg Part 1 | AZD3293 150 mg Part 1 | AZD3293 15 mg Part 2 | AZD3293 50 mg Part 2 | Placebo Part 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/6 | 0/6 | 2/6 | 2/6 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Part 1 (N=6) | AZD3293 15 mg Part 1 (N=6) | AZD3293 50 mg Part 1 (N=6) | AZD3293 150 mg Part 1 (N=6) | AZD3293 15 mg Part 2 (N=6) | AZD3293 50 mg Part 2 (N=6) | Placebo Part 2 (N=4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nasopharengitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days